CLINICAL TRIAL: NCT00784888
Title: A Non-Interventional Study Evaluating The Effects Of Aromatase Inhibitor Treatment After 2-3 Years Tamoxifen - As Adjuvant Endocrine Therapy - On Quality Of Life And Safety In Endocrine Responsive Early Stage Postmenopausal Breast Cancer Patients
Brief Title: Research Of Quality Of Life And Safety Outcomes Of Postmenopausal Breast Cancer Patients Switching From Tamoxifen Therapy To Aromatase Inhibitor Therapy
Acronym: TAMARA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5991087
Record Dates: First submitted 2008-10-31; First posted 2008-11-04 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Breast Neoplasms
Keywords: aromatase inhibitor; quality of life; safety; postmenopausal breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aromatase inhibitors: Early stage postmenopausal breast cancer patients under tamoxifen treatment who are switching to aromatase inhibitor treatment
  Interventions: Other: Aromatase inhibitors

INTERVENTIONS:
Other: Aromatase inhibitors — non-interventional study

SUMMARY:
The purpose of this study is to follow safety and quality of life outcomes on patients switching from tamoxifen therapy to aromatase inhibitor therapy.

DETAILED DESCRIPTION:
Group of patients using the same aromatase inhibitor

ELIGIBILITY:
Inclusion Criteria:

Patients with endocrine responsive early stage postmenopausal breast cancer. Patients who received tamoxifen for 2-3 years as adjuvant endocrine therapy. Patients who were approved to switch to aromatase inhibitor treatment during the patient recruitment period.

Patients who were informed about the study and accepted to participate.

Exclusion Criteria:

Patients having a psychological disorder which will prevent their understanding of questionnaires used for evaluation of quality of life and / or patients who are illiterate.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endocrine responsive early stage postmenopausal breast cancer. Patients who received tamoxifen for 2-3 years as adjuvant endocrine therapy. Patients who were approved to switch to aromatase inhibitor treatment during the patient recruitment period.
  Patients who were informed about the study and accepted to participate.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the quality of life of patients with early stage postmenopausal breast cancer using aromatase inhibitor following 2-3 years of tamoxifen treatment (switch) | 2 years

SECONDARY OUTCOMES:
To evaluate patients with early stage postmenopausal breast cancer using aromatase inhibitor following 2-3 years of tamoxifen treatment (switch) in terms of side effects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Turkey (Türkiye) (12):
  - Pfizer Investigational Site, Adana
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Bursa
  - Pfizer Investigational Site, Denizli
  - Pfizer Investigational Site, Edirne
  - Pfizer Investigational Site, Erzurum
  - Pfizer Investigational Site, Gaziantep
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, Kocaeli
  - Pfizer Investigational Site, Malatya
  - Pfizer Investigational Site, Trabzon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991087&StudyName=Research%20Of%20Quality%20Of%20Life%20And%20Safety%20Outcomes%20Of%20Postmenopausal%20Breast%20Cancer%20Patients%20Switching%20From%20Tamoxifen%20Therapy%20To%20Aromatase%20I